CLINICAL TRIAL: NCT07222514
Title: Feasibility and Safety of Single-Port Robotic-Assisted DIEP Flap Harvest for Breast Reconstruction: A Prospective Evaluation
Brief Title: Feasibility and Safety of Single-Port Robotic-Assisted Deep Inferior Epigastric Pedicle Flap Harvest
Acronym: (DIEP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, Galen Perdikis, Chair and Professor, Department of Plastic Surgery, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 250009
Record Dates: First submitted 2025-09-09; First posted 2025-10-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: DIEP Flap Breast Reconstruction
Keywords: DIEP flap breast reconstruction; Robotic Surgery; Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Robotic Assisted DIEP Breast Reconstruction (Experimental): This group consists of patients receiving the investigative procedure - robotic assisted DIEP flap harvest for breast reconstruction.
  Interventions: Device: Single-Port Robotic System

INTERVENTIONS:
Device: Single-Port Robotic System — Utilizing the Single-Port robotic system for DIEP flap harvest has been previously described, but only in a small pilot study. The investigators plan to demonstrate the feasibility and safety of this approach on a larger cohort of patients.

SUMMARY:
The primary aim of this study is to evaluate the feasibility of single-port robotic surgery for DIEP flap breast reconstruction. The investigators will also investigate complications of the procedure, incision length, flap success rate, post operative pain, vascular pedicle length and caliber, and VMP-B score (quality of life/satisfaction of breast procedures survey).

DETAILED DESCRIPTION:
This project will be conducted at Vanderbilt University Medical Center. Patients scheduled for a DIEP flap procedure will be recruited through screening of the electronic medical records (EMR) to evaluate eligibility based on pre-established inclusion and exclusion criteria. Eligible patients will be invited to participate in a preoperative consultation, during which they will receive detailed information about the study, including the surgical techniques, potential risks, and benefits. Written informed consent will be obtained from those who agree to participate.

Baseline data available in the medical records as part of their clinical care, including patient demographics, medical history, imaging, pictures, pain and quality-of-life metrics, will also be collected.

On the day of surgery, patients will undergo standard preoperative preparations. The procedure will involve robotic-assisted DIEP flap harvest using single-port access, followed by flap transfer and microsurgical anastomosis. Post-surgical donor site closure will employ techniques to minimize morbidity. Key intraoperative data, such as operative time and complications, will be recorded.

Patient Electronic Medical Records (EMR) will be accessed by research personnel to monitor patients who elect to have the proposed procedure. Postoperative monitoring will focus on flap viability and patient recovery during the hospital stay and subsequent follow-ups. Assessments will include complications, donor site integrity, pain levels, and patient-reported outcomes. Follow-up visits will evaluate both short- and long-term outcomes, including satisfaction and quality of life, providing comprehensive data for the study's primary and secondary aims.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Candidates for unilateral or bilateral breast reconstruction using a DIEP flap.
* No contraindications for general anesthesia or robotic surgery.
* Patients with adequate abdominal donor tissue for DIEP flap harvest.

Exclusion Criteria:

* History of prior abdominal surgery that significantly compromises perforator vessel integrity.
* Pregnant woman.
* Prisoners.
* BMI > 35, as measured during the preoperative evaluation.
* Presence of comorbidities that contraindicate elective surgery.
* Active cancer other than breast cancer at the time of evaluation.
* Active metastatic disease confirmed via imaging or biopsy.
* Inability to comply with follow-up visits.
* The research team decides to exclude the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing DIEP flap breast construction using a single port robotic system | From enrollment to the end of the procedure.
  This will be "Yes" if the following are true of the procedure: completed pedicle dissection using the robotic system, adequate pedicle dissected, and no intraoperative complication requiring conversion to the open approach.

SECONDARY OUTCOMES:
Complication Rates | Through study completion, an average of 1 year.
  Intraoperative and postoperative complications. Including, but not limited to: flap failure, internal structure injuries, deep venous thrombosis, etc.
Fascial Incision Length | Through study completion, an average of 1 year.
  Measurement of the fascial incision length and prevalence of abdominal herniation or bulging through the incision.
Flap Success Rate | From procedure to 7 days post operation.
  We define flap success rate as survival of the flap without loss of viability through a specified time window.
Operative Time | From procedure start to procedure completion.
  The time interval between first skin incision to skin closure of the patient.
Pain Level | From procedure to postoperative day (POD) 1, 2, 3, 7, 14, and 30.
  The patient level of pain on a scale of 1 (no pain) to 10 (extreme pain).
Vascular Pedicle Length | During the operative procedure (approximately 6 - 10 hours, intraoperative measurement)
  The pedicle length used for anastomosis will be measured intraoperatively, reported in mm.
Vanderbilt Mini Patient Reported Outcome - Breast (VMP-B) Score | From enrollment to 12 months post operation. Surveys will be distributed preoperatively and at postoperative follow up intervals (2 weeks, 6 weeks, 3 months, 6 months, and 12 months).
  The investigators will collect patient VMP-B (a validated patient reported outcome) scores to assess patient well being and satisfaction with their procedure. Items (16 total) are scored on a 5-point Likert scale, scores range from 16 (worst) to 80 (best).
Pain Management | From procedure to postoperative day (POD) 1, 2, 3, 7, 14, and 30.
  The investigators will record what analgesics are used to control patient pain.
Vascular Pedicle Caliber | During the operative procedure (approximately 6 - 10 hours, intraoperative measurement)
  The pedicle caliber used for anastomosis will be measured intraoperatively, reported in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Galen Perdiks, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
As this is a feasibility study - there is no indication to share individual participant data.

REFERENCES:
- [Background] Roy N, Alessandro CJ, Ibelli TJ, Akhavan AA, Sharaf JM, Rabinovitch D, Henderson PW, Yao A. The Expanding Utility of Robotic-Assisted Flap Harvest in Autologous Breast Reconstruction: A Systematic Review. J Clin Med. 2023 Jul 27;12(15):4951. doi: 10.3390/jcm12154951. PMID 37568353
- [Background] Tsai CY, Kim BS, Kuo WL, Liu KH, Chang TN, Cheong DC, Huang JJ. Novel Port Placement in Robot-Assisted DIEP Flap Harvest Improves Visibility and Bilateral DIEP Access: Early Controlled Cohort Study. Plast Reconstr Surg. 2023 Oct 1;152(4):590e-595e. doi: 10.1097/PRS.0000000000010470. Epub 2023 Mar 30. PMID 36995211
- [Background] Lee MJ, Won J, Song SY, Park HS, Kim JY, Shin HJ, Kwon YI, Lee DW, Kim NY. Clinical outcomes following robotic versus conventional DIEP flap in breast reconstruction: A retrospective matched study. Front Oncol. 2022 Sep 14;12:989231. doi: 10.3389/fonc.2022.989231. eCollection 2022. PMID 36185209
- [Background] Choi JH, Song SY, Park HS, Kim CH, Kim JY, Lew DH, Roh TS, Lee DW. Robotic DIEP Flap Harvest through a Totally Extraperitoneal Approach Using a Single-Port Surgical Robotic System. Plast Reconstr Surg. 2021 Aug 1;148(2):304-307. doi: 10.1097/PRS.0000000000008181. PMID 34398082